CLINICAL TRIAL: NCT05429632
Title: Randomized, Double-blind, Placebo-controlled, Multi-center Phase III Study to Evaluate the Efficacy and Safety of Mocravimod as Adjunctive and Maintenance Treatment in Adult AML Patients Undergoing Allogeneic HCT
Brief Title: Mocravimod as Adjunctive and Maintenance Treatment in AML Patients Undergoing Allo-HCT
Acronym: MO-TRANS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Priothera SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Priothera SAS
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, randomized, double-blind, placebo-controlled, and 3-arm parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 3mg mocravimod arm (Experimental): 3 mg of mocravimod orally once per day for 12 months
  Interventions: Drug: mocravimod
- 1mg mocravimod arm (Experimental): 1 mg of mocravimod orally once per day for 12 months
  Interventions: Drug: mocravimod
- Placebo arm (Placebo Comparator): placebo orally once per day for 12 months
  Interventions: Drug: mocravimod

INTERVENTIONS:
Drug: mocravimod — S1PR modulator

SUMMARY:
This is a multi-center, randomized, double-blinded, placebo controlled trial.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of mocravimod as an adjunctive and maintenance treatment in adult acute myeloid leukemia (AML) patients undergoing allogeneic hematopoietic cell transplantation (HCT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML (excluding acute promyelocytic leukemia) according to the WHO 2022 classification of AML and related precursor neoplasm, including AML with myelodysplasia-related gene mutations
* European Leukemia Net (ELN) high-risk or intermediate-risk AML in CR1, or AML of any risk in CR2, [CRi] is also allowable
* Planned allogeneic HCT from fully matched related or unrelated donor with no more than 1 antigen mismatch or planned use of haploidentical donor using PBSC graft
* Any conditioning regimen with a Transplant Conditioning Score (TCI) ≥ 1.5
* Planned use of TAC-based GvHD prophylaxis
* age ≥ 18 years and ≤ 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Use of CsA, anti-thymocyte globulin (ATG), alemtuzumab, abatacept for GvHD prophylaxis
* Diagnosis of macular edema during screening
* Cardiac/pulmonary/hepatic/renal dysfunction
* Hepatic dysfunction as defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN); or total bilirubin > 1.5 mg/dL
* Renal dysfunction with estimated creatinine clearance < 45 mL/min by the Cockcroft-Gault formula

  * Diabetes mellitus
  * History or presence of uveitis at screening
  * History or diagnosis of macular edema

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | 12 months
  To compare the efficacy of mocravimod to that of placebo

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  To compare mocravimod's effect on overall survival (OS) to that of placebo

CONTACTS AND LOCATIONS:
Overall Officials: Marcos DeLima, MD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (108):
- United States (21):
  - University of Alabama Hospital (UAB Hospital), Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope Comprehensive Cancer Center - Duarte, Duarte, California
  - University of California Los Angeles (UCLA) - David Geffen School of Medicine, Los Angeles, California
  - UCHealth Cancer Care - Anschutz Medical Campus - University of Colorado Cancer Center, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University - Winship Cancer Institute (WCI), Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Ochsner Medical Center (OMC) - New Orleans, New Orleans, Louisiana
  - University of Maryland Medical Center (UMMC), Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Spectrum Health Medical Group (SHMG) - Blood & Marrow Transplant - Adult (BMT), Grand Rapids, Michigan
  - University of Rochester Medical Center (URMC), Rochester, New York
  - Stony Brook University (SBU) - Cancer Center, Stony Brook, New York
  - University of Cincinnati Medical Center (University Hospital), Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center (OSUCCC), Cleveland, Ohio
  - Oregon Health & Science University (OHSU) - Knight Cancer Institute, Portland, Oregon
  - University of Pennsylvania - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
- Argentina (4):
  - Hospital El Cruce - Dr. Nestor Kirchner, Buenos Aires
  - Centro de Educacion Medica E Investigacines Clinicas Norberto Quirno CEMIC, Buenos Aires
  - Sanatorio Allende (SA) - Nueva Cordoba, Córdoba
  - Hospital Italiano La Plata, La Plata
- Brazil (7):
  - CEPON - Centro de Pesquisas Oncologicas, Florianópolis, Santa Catarina
  - Hospital Erasto Gaertner, Curicica
  - Hospital Alemao Oswaldo Cruz (HAOC), São Paulo
  - Universidade de Sao Paulo (USP) - Hospital das Clinicas da Faculdade de Medicina (HCFMUSP), São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Unicamp, São Paulo
  - Hospital Amaral Carvalho, São Paulo
- France (8):
  - Centre Hospitalier Universitaire (CHU) Angers, Angers
  - Centre Hospitalier Regional Universitaire (CHRU) de Lille - Hopital Claude Huriez -, Lille
  - Centre Hospitalier Lyon-Sud, Lyon
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Hospital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse
  - Centre de Lutte Contre le Cancer (CLCC) - Institut Gustave-Roussy, Villejuif
- Germany (4):
  - Universitätsklinikum Halle, Halle
  - Universitaetsklinikum Jena - Klinik fuer Innere Medizin II, Jena
  - University of Leipzig Medical Center, Leipzig
  - LMU Klinikum Grosshadern Klinikum der Universitaet Muenchen, Munich
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (12):
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli, Reggio Calabria, Calabria
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale Casa Sollievo della Sofferenza (CSS), San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo Alessandria, Alessandria
  - Azienda Sanitaria Locale 13 - Ospedale "C. e G. Mazzoni"- Ascoli Piceno, Ascoli Piceno
  - Azienda Sanitaria Localedella provincia di Brindisi -, Brindisi
  - Universita degli Studi di Firenze - Azienda Ospedaliero-Universitaria Careggi (AOUC) LAB TMO, Florence
  - Ospedale Vito Fazzi Lecce, Lecce
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera San Gerardo - Monza, Monza
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Japan (15):
  - Anjo-kosei Hospital, Anjo-shi, Aichi-ken
  - Japanese Red Cross Nagoya Daiichi Hospital (First Hospital), Nagoya, Aichi-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Jichi Medical University (JMU) Hospital, Shimotsuke-shi, Tochigi
  - Kyushu University Hospital,, Fukuoka
  - Hiroshima Red Cross Hospital & Atomic-Bomb Survivors Hospital, Hiroshima
  - Kobe City Medical Center General Hospital, Kobe
  - Kyoto University Hospital, Kōtoku
  - Ehime Prefectural Centeral Hospital, Ehime, Matsuyama
  - Okayama University Hospital, Okayama
  - Jichi Medical University Saitama Medical Center, Saitama
  - Hokkaido University Hospital, Sapporo
  - Tokyo Metropolitan Cancer and infection Disese Center Komagome Hospital, Tokyo
  - Oita University (OU) Hospital, Yufu
- Poland (5):
  - Sp Zoz Szpital Uniwersytecki W Krakowie, Krakow, Aichi-Ken
  - Slaski Uniwersytet Medyczny (SUM) w Katowicach - Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mieleckiego (SPSKM) - Slaskie Centrum Hematologii I Transplantacji Szpiku, Katowice, Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne (UCK), Gdansk
  - Apteka NSSU, Krakow
  - Centralny Szpital Kliniczny Apteka Szpitalna, Warsaw
- Romania (3):
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Institutul Regional de Oncologie Iasi, - Haematology Department, Iași
- Spain (10):
  - Hospital Universitari Vall d'Hebron - Institut de Recerca (VHIR), Barcelona
  - Institut Catala d'Oncologia (ICO), Barcelona
  - Institut Catala d'Oncologia (ICO) - Hospital Universitari Germans Trias i Pujol (HUGTP) Location, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Gran Canaria "", Las Palmas de Gran Canaria
  - Hospital De La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico Universitario - Universidad de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe, Valencia
- Universitaetsspital Basel, Basel, Switzerland
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital (NTUH), Taipei
  - National Taiwan University Cancer Center, Taipei
- United Kingdom (10):
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital of Wales, Cardiff, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - University College Hospital,, London
  - Imperial College, London, London
  - Manchester Royal Infirmary;Manchester University, Manchester
  - Newcastle Upon Tyne Hospitals Norhtern Center for Cancer Care, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals, Oxford
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No